CLINICAL TRIAL: NCT01596699
Title: A Pilot Trial of Clofarabine Added to Standard Busulfan and Fludarabine for Conditioning Prior to Allogeneic Hematopoietic Cell Transplantation
Brief Title: Pilot Trial of Clofarabine Added to Standard Busulfan and Fludarabine for Conditioning Prior to Allogeneic Hematopoietic Cell Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Triggering of futility rule; Interim analysis suggested no statistical superiority over historic controls
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110819; NCI-2012-00800 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2012-05-07; First posted 2012-05-11 (Estimated); Results first posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Myeloid Malignancy; Bone Marrow Failure Syndrome; Transfusion-dependent Red Blood Cell (RBC) Defect; Congenital Immunodeficiency; Metabolic Disease; Severe Immune Dysregulation
Keywords: conditioning; allogeneic; hematopoietic; cell; transplantation; HCT
MeSH Terms: conditions — Bone Marrow Failure Disorders; Metabolic Diseases | interventions — Alemtuzumab; Busulfan; fludarabine; fludarabine phosphate; Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patients with Myeloid Malignancies (Experimental)
  Interventions: Drug: Busulfan; Drug: Fludarabine; Drug: Clofarabine
- Patients with Non-Malignancies (Experimental)
  Interventions: Drug: Alemtuzumab; Drug: Busulfan; Drug: Fludarabine; Drug: Clofarabine

INTERVENTIONS:
Drug: Alemtuzumab — 0.5 mg/kg (max 15 mg or max 6 mg), IV, Day -12 to Day -10 pre-HCT
  Other Names: Campath
  Arms: Patients with Non-Malignancies
Drug: Busulfan — 0.8 mg/kg/dose q6hrs or 1.1 mg/kg/dose q6hrs, IV, Day -9 to Day -6 pre-HCT
  Other Names: Busulfex
Drug: Fludarabine — 40 mg/m2 or 1.33 mg/kg, IV, Day -5 to Day -2 pre-HCT
  Other Names: Fludara
Drug: Clofarabine — 10 mg/m2 or 0.33 mg/kg, IV, Day -5 to Day -2 pre-HCT
  Other Names: Clolar

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, the addition of clofarabine, a new chemotherapy agent, to a standard busulfan and fludarabine conditioning treatment has. The study will also look at what causes some people to have high drug levels of these medications in their body compared to other people that may have low drug levels even if they all receive the same dose of medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 3 months and ≤30 years of age.
* Stratum A: Non-Malignant Diseases, including:

  * Bone Marrow Failure Syndromes
  * Hemoglobinopathies or transfusion-dependent red blood cell (RBC) defects
  * Congenital Immunodeficiencies
  * Metabolic Diseases known to be treatable with Hematopoietic cell transplantation (HCT) (e.g. Hurler's)
  * Other Bone Marrow Stem Cell Defects (e.g. Osteopetrosis)
  * Severe Immune Dysregulation / Autoimmune Syndromes with at least transient prior response to immunosuppressive therapy
* Stratum B: Myeloid Malignancies, including:

  * acute myeloid leukemia (AML), in greater than first clinical remission, or in CR1 but with detectable disease (≥0.1% Blasts by minimal residual disease (MRD) or Flow, or Positive Cytogenetics), or in CR1 but with a matched sibling Umbilical cord blood (UCB) donor.
  * Myelodysplastic syndromes (MDS)
  * Juvenile myelomonocytic leukemia (JMML)
  * Chronic myeloid leukemia (CML), with detectable disease by polymerase chain reaction (PCR)
* Patients must have a suitable donor based on the University of California, San Francisco (UCSF) Pediatric Bone Marrow Transplant (BMT) standard operating procedures (SOP). 10/10 (HLA-A, -B, -C, -DR, -DQ) matching will be done for related and adult unrelated donors; 8/8 (HLA-A, -B, -C, -DR) for umbilical cord blood donors. Patients with non-malignant diseases will generally be eligible only if they have a mismatched donor, or an accepted clinical reason to be considered high-risk for rejection.
* Liver transaminases (aspartate aminotransferase (AST)/alanine aminotransferase (ALT)) and Direct Bilirubin less than twice the upper limit of normal within 2 weeks of admission.
* Cardiac Shortening Fraction ≥27% within 4 weeks of admission.
* Creatinine clearance by Schwartz formula, glomerular filtration rate (GFR) or 24 hr urine collection ≥50 cc/min/1.73 m2, within 4 weeks of admission.
* Pulmonary diffusion capacity ≥50% of predicted corrected for anemia/lung volume within 4 weeks of admission. If unable to do Pulmonary function testing(PFTs), then no active lung disease by chest x-ray (CXR) and/or oxygen (O2) Saturation ≥90% on room air.

Exclusion Criteria:

* Fanconi Anemia
* Dyskeratosis Congenita
* A known syndrome with increased sensitivity to radiation or alkylating agents
* Severe Combined Immunodeficiency Disease eligible for a non-myeloablative HCT Trial
* A mismatched donor for whom ex vivo T-cell depletion of the donor stem cells is planned

Ages: 3 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2012-05-24 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C Dvorak, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Stratum A: Patients With Non-Malignancies: Alemtuzumab: 0.5 mg/kg (max 15 mg or max 6 mg), IV, Day -12 to Day -10 pre-Hematopoietic cell transplantation (HCT)
  Busulfan: 0.8 mg/kg/dose q6hrs or 1.1 mg/kg/dose q6hrs, IV, Day -9 to Day -6 pre-HCT
  Fludarabine: 40 mg/m2 or 1.33 mg/kg, IV, Day -5 to Day -2 pre-HCT
  Clofarabine: 10 mg/m2 or 0.33 mg/kg, IV, Day -5 to Day -2 pre-HCT
- Stratum B: Patients With Myeloid Malignancies: Busulfan: 0.8 mg/kg/dose q6hrs or 1.1 mg/kg/dose q6hrs, IV, Day -9 to Day -6 pre-HCT
  Fludarabine: 40 mg/m2 or 1.33 mg/kg, IV, Day -5 to Day -2 pre-HCT
  Clofarabine: 10 mg/m2 or 0.33 mg/kg, IV, Day -5 to Day -2 pre-HCT
Period: Overall Study
Arm/Group | Stratum A: Patients With Non-Malignancies | Stratum B: Patients With Myeloid Malignancies
Started | 10 | 6
Completed | 10 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Stratum A: Patients With Non-Malignancies: Alemtuzumab: 0.5 mg/kg (max 15 mg or max 6 mg), IV, Day -12 to Day -10 pre-HCT
  Busulfan: 0.8 mg/kg/dose q6hrs or 1.1 mg/kg/dose q6hrs, IV, Day -9 to Day -6 pre-HCT
  Fludarabine: 40 mg/m2 or 1.33 mg/kg, IV, Day -5 to Day -2 pre-HCT
  Clofarabine: 10 mg/m2 or 0.33 mg/kg, IV, Day -5 to Day -2 pre-HCT
- Total: Total of all reporting groups
Arm/Group | Stratum A: Patients With Non-Malignancies | Stratum B: Patients With Myeloid Malignancies | Total
Number analyzed (Participants) | 10 | 6 | 16
Age, Customized [Count of Participants; unit: Participants]
  0-9 years old | 10 | 6 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 7 | 3 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Related Adverse Events as a Measure of Safety and Tolerability
Description: Severe Toxicity will be defined as death or Grade IV by NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 pulmonary or hepatic failure (including moderate veno-occlusive disease(VOD) related to the transplant conditioning regimen within 100 days post-HCT. VOD will be defined by standard criteria. Patients must have Bilirubin >2.0 plus Hepatomegaly and/or Right upper quadrant (RUQ) pain plus Weight gain >5%.
Time Frame: Up to 5 years on average
Measure: Number; unit: participants
Arm/Group | Stratum A: Patients With Non-Malignancies | Stratum B: Patients With Myeloid Malignancies
Number analyzed (Participants) | 10 | 6
participants
  Death | 1 | 0
  Veno-occlusive disease(VOD) | 1 | 1

2. Secondary Outcome: Engraftment Rate of Patients With Non-malignant Diseases (Stratum A)
Description: Engraftment will be defined as the development of an Absolute Neutrophil Count (ANC) >500 for 3 consecutive days plus donor CD14/15 cells >70%. The engraftment rate in the population used for historical control is 40%. If 3 patients in Stratum A experience graft rejection, this stratum will close early for failing to achieve superior engraftment compared to standard-of-care.
Time Frame: Participants will have engraftment blood studies starting approximately Day 30 post hematopoietic stem cell transplant and then monthly until stable. Average study participation is approximately 5 years.
Population: Three patients in Stratum A experienced graft rejection which met the criteria for failing to achieve superior engraftment compared to standard-of-care. One patient was not evaluable.
Measure: Number; unit: percentage of participants
Arm/Group | Stratum A: Patients With Non-Malignancies
Number analyzed (Participants) | 9
percentage of participants | 66.67

3. Secondary Outcome: Mixed-donor Chimerism Rate of Patients With High-risk Myeloid Malignancies (Stratum B)
Description: Full-donor chimerism will be defined by as ≥99% donor cells by Short Tandem Repeat (STR) analysis in all cell lines (CD3, CD14/15, and CD19) in peripheral blood. The historic control for Stratum B was determined using the 20 patients who were transplanted from 2005 - 2010 with Busulfan (BU)-based regimens and who retrospectively would have been eligible for the current trial. Of these 20 patients, at 100 days post-HCT, only 8 (40%) patients had full-donor chimerism. If 5 patients in Stratum B experienced mixed-donor chimerism at Day 100, we will close this stratum early for failing to achieve superior donor cell engraftment compared to standard-of-care.
Time Frame: Participants will have peripheral blood chimerism assessed at Day 100 post hematopoietic stem cell transplant and then monthly until stable.
Measure: Number; unit: percentage of participants
Arm/Group | Stratum B: Patients With Myeloid Malignancies
Number analyzed (Participants) | 6
percentage of participants | 66.67

4. Secondary Outcome: Serum Concentrations and Potential for Drug-drug Interaction of Fludarabine and Clofarabine
Description: Fludarabine and clofarabine drug levels and potential covariates influencing drug exposure such as renal function and genetic variants involved in drug metabolism, distribution, and activation will be analyzed using standard population pharmacokinetic methods using non-linear mixed effects modeling (NONMEM) software
Time Frame: Pharmacokinetics (PK) blood sampling Days -5 to -2 pre-hematopoietic stem cell transplant.
Population: PK Data not collected
Arm/Group | Stratum A: Patients With Non-Malignancies | Stratum B: Patients With Myeloid Malignancies
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: Bone Marrow Transplant (BMT) patients have a large number of toxicities as an expected part of the intervention. Some traditional adverse events are an intended part of the conditioning and therefore not considered an unexpected toxicity as part of the treatment regimen. All of the reported febrile neutropenia, anemia, and mucositis events were anticipated as part of bone marrow transplant.
Arm/Group | Stratum A: Patients With Non-Malignancies | Stratum B: Patients With Myeloid Malignancies
All-Cause Mortality (participants affected / at risk) | 1/10 | 6/6
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/6
Other Adverse Events (participants affected / at risk) | 10/10 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum A: Patients With Non-Malignancies (N=10) | Stratum B: Patients With Myeloid Malignancies (N=6)
Veno-occlusive disease (VOD) (General disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum A: Patients With Non-Malignancies (N=10) | Stratum B: Patients With Myeloid Malignancies (N=6)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 10 (10) | 6 (6)
Anemia (Blood and lymphatic system disorders) | 10 (10) | 6 (6)
Mucositis oral (Gastrointestinal disorders) | 10 (10) | 6 (6)
Lung Infection (Infections and infestations) | 0 (0) | 1 (1)
Lymph Gland Infection (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study closed prior to completion. Interim analysis suggested treatments would not demonstrate statistical superiority over historic controls.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2013-06-07): https://cdn.clinicaltrials.gov/large-docs/99/NCT01596699/Prot_SAP_000.pdf
  • Informed Consent Form: Minor-Parental (2014-04-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT01596699/ICF_001.pdf
  • Informed Consent Form: Assent (Ages 7-12) (2014-04-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT01596699/ICF_002.pdf
  • Informed Consent Form: Adult Adolescent (2014-04-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT01596699/ICF_003.pdf